CLINICAL TRIAL: NCT04143490
Title: The Effects of Exercise Intensity on Gastrointestinal Function and Inflammatory Markers in Patients With Ulcerative Colitis
Brief Title: Effects of Exercise in Patients With Ulcerative Colitis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid-19
Sponsor: Manchester Metropolitan University (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Adora Yau, Lecturer, Manchester Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ExerciseUC-2019
Record Dates: First submitted 2019-10-15; First posted 2019-10-29 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease; Exercise; Gastric emptying rate; Inflammatory markers; Gastrointestinal integrity
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single experimental trial with a UC patient group and an age and gender matched healthy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC Patients (Experimental): Patient group
  Interventions: Other: Exercise
- Healthy controls (Active Comparator): Control group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 60 minutes of continuous exercise at 65% VO2peak and drink ingestion

SUMMARY:
The aim of this study is to investigate the effects of moderate to high intensity exercise on gut function and inflammatory markers in patients with Ulcerative Colitis (UC), and to compare them with individuals of matched age who do not suffer from Inflammatory Bowel Disease. Participants will be asked to complete 60 minutes of continuous cycling at a moderate to high intensity followed by a three hour recovery period. Gastrointestinal function will be measured using a non-invasive breath test. Blood samples will be collected at multiple time-points during the visit and these samples will be measured for markers of immune function and intestinal integrity.

DETAILED DESCRIPTION:
There is limited research on the effect of exercise on patients with Ulcerative Colitis. The aim of this investigation is to study the acute effects of moderate to high intensity exercise on gut function in patients with Ulcerative Colitis and to compare them with individuals of matched age who do not suffer from Inflammatory Bowel Disease.

Patients in remission from disease activity and age and gender matched healthy control participants will be recruited from the general population. Participants will attend the laboratory on two occasions. The first visit will last approximately one hour and will include an exercise test to determine peak oxygen uptake capacity (VO2peak) which is an indicator of cardiorespiratory fitness. The second visit will last for approximately four and a half hours and will consist of a 60 minute continuous cycle on a stationary cycle ergometer at an intensity of 65% VO2peak followed by a recovery period. Gastric emptying rate of a commercially available sports drink will be measured and blood samples will be collected at regular time-points throughout the visit and analysed for concentrations of inflammatory markers and intestinal integrity/function.

ELIGIBILITY:
Inclusion Criteria:

For ulcerative colitis patients;

* Currently in remission of disease (asymptomatic at time of experiment)
* Less than 3 periods of disease activity (periods of symptomatic activity) in the last 12 months
* No history of surgery to alleviate condition severity
* Taking regular standard medication for control of condition
* Adult less than 50 years due to effects of exercise in older age
* Non-smokers
* Regular exercisers (determined via verbal discussion)

For healthy controls;

* No history of disease (as assessed by standard medical screening questionnaire)
* Adult less than 50 years due to effects of exercise in older age
* Non-smokers
* Regular exercisers (determined via verbal discussion)

Exclusion Criteria:

For ulcerative colitis patients;

* Currently in active period of disease (symptomatic at time of experiment)
* More than 3 periods of disease activity (periods of symptomatic activity) in the last 12 months
* History of surgery to alleviate condition severity
* Taking non-standard medication for control of condition
* Adult more than 50 years of age
* Under 18 years of age
* Smokers
* Sedentary or not regularly physically active (determined via verbal discussion)

For healthy controls;

* History of disease (as assessed by standard medical screening questionnaire)
* Adult more than 50 years of age
* Under 18 years of age
* Smokers
* Sedentary or not regularly physically active (determined via verbal discussion)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory markers or hormones | 6 blood samples collected at baseline, 30 minutes of exercise (mid exercise), immediately post exercise bout, then every 60 minutes post exercise for 3 hours
  Circulating concentrations of Interleukin-6, Tumor Necrosis Factor-alpha, C-reactive protein, glucagon like peptide 2
Area under the circulating concentration versus time curve (AUC) of inflammatory markers or hormones | 4.5 hours
  Responses of Interleukin-6, Tumor Necrosis Factor-alpha, C-reactive protein, glucagon like peptide 2
Change in intestinal epithelial damage and permeability markers | 6 blood samples collected at baseline, 30 minutes of exercise (mid exercise), immediately post exercise bout, then every 60 minutes post exercise for 3 hours
  Circulating concentrations of intestinal fatty acid binding protein and claudin-3
Area under the circulating concentration versus time curve (AUC) of intestinal epithelial damage and permeability markers | 4.5 hours
  Responses of intestinal fatty acid binding protein and claudin-3
Change in exercise induced endotoxaemia markers | 6 blood samples collected at baseline, 30 minutes of exercise (mid exercise), immediately post exercise bout, then every 60 minutes post exercise for 3 hours
  Circulating concentrations of plasma lipopolysaccharide
Area under the circulating concentration versus time curve (AUC) of exercise induced endotoxaemia markers | 4.5 hours
  Response of plasma lipopolysaccharide
Gastric emptying rate half time and time of maximal emptying rate | 2 hours after ingestion of drink
  Emptying rate of a commercially available sports drink from the stomach using the 13C breath test method
Change in ratio of 13C/12C in breath samples | 9 breath samples collected at baseline, then every 15 minutes after ingestion for 2 hours
  Gastric emptying profile of a commercially available sports drink from the stomach using the 13C breath test method

SECONDARY OUTCOMES:
Incidence and severity of gastrointestinal symptoms | Immediately post-exercise bout and 3 hours post exercise.
  10-point rating scale for gastrointestinal symptoms (Visual Analogue Scale modified). 19 item questionnaire with 5 subcategories (Overall gut discomfort, total gastrointestinal symptoms, upper gastrointestinal symptoms, lower gastrointestinal symptoms and other gastrointestinal symptoms). Scores for each item ranging from 0 (no symptom) to 10 (extremely severe symptoms causing exercise reduction, stopping, or complete withdrawal). Higher scores represent higher severity of symptoms.
Heart rate response | Every 5 minutes during 60 minute cycle
  Heart rate telemetry
Disparity of subjective exertion and objective cardiorespiratory parameters | Every minute during the peak oxygen uptake test that typically lasts between 8-12 minutes
  Regression of ratings of perceived exertion (RPE; Borg scale, minimum value 6 representing no exertion, maximum value 20 representing maximal exertion. Higher scores represent higher perceived exertion) and cardiopulmonary exercise testing variables of oxygen uptake, carbon dioxide expiration, ventilatory threshold, volume of air expired, and tidal volume (all parameters measured in L/min).
Disparity of subjective exertion and objective heart rate | Every minute during the peak oxygen uptake test that typically lasts between 8-12 minutes
  Regression of ratings of perceived exertion (RPE; Borg scale, minimum value 6 representing no exertion, maximum value 20 representing maximal exertion. Higher scores represent higher perceived exertion) and heart rate measured by telemetry
Disparity of subjective exertion and breathing frequency | Every minute during the peak oxygen uptake test that typically lasts between 8-12 minutes
  Regression of ratings of perceived exertion (RPE; Borg scale, minimum value 6 representing no exertion, maximum value 20 representing maximal exertion. Higher scores represent higher perceived exertion) and number of breaths per minute
Disparity of subjective exertion and oxygen pulse | Every minute during the peak oxygen uptake test that typically lasts between 8-12 minutes
  Regression of ratings of perceived exertion (RPE; Borg scale, minimum value 6 representing no exertion, maximum value 20 representing maximal exertion. Higher scores represent higher perceived exertion) and oxygen pulse calculated by dividing oxygen uptake by heart rate.
Disparity of subjective exertion and respiratory exchange ratio | Every minute during the peak oxygen uptake test that typically lasts between 8-12 minutes
  Regression of ratings of perceived exertion (RPE; Borg scale, minimum value 6 representing no exertion, maximum value 20 representing maximal exertion. Higher scores represent higher perceived exertion) and respiratory exchange ratio calculated by dividing carbon dioxide production by oxygen uptake.
Disparity of subjective exertion and ventilatory efficiency | Every minute during the peak oxygen uptake test that typically lasts between 8-12 minutes
  Regression of ratings of perceived exertion (RPE; Borg scale, minimum value 6 representing no exertion, maximum value 20 representing maximal exertion. Higher scores represent higher perceived exertion) and minute ventilation/carbon dioxide slope (VE/VCO2 slope).
Subjective physical activity levels | Prior to experimental trial
  International Physical Activity Questionnaire (IPAQ). Answers to questions (time spent completing different physical activities) converted to Metabolic Equivalent (METs) hours per week. Minimum value of zero, no limit to maximum. Higher MET values indicate higher physical activity levels.
Attitudes and beliefs towards physical activity | Prior to experimental trial
  Barriers to Physical Activity Questionnaire. 21 item questionnaire, each question rated from 0 (very unlikely) to 3 (very likely). Each item belongs to one of 7 categories relating to barriers to physical activity. Score totals greater than 5 indicate the category as being a significant barrier.
Subjective health related quality of life: RAND 36-Item Short Form Health Survey (SF-36) | Prior to experimental trial
  RAND 36-Item Short Form Health Survey (SF-36). 36-item questionnaire covering 8 concepts; physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions, plus single item providing an indication of perceived change in health. Scores ranging from 0 to 100 for each concept with 100 indicating good health and 0 being poor health.

CONTACTS AND LOCATIONS:
Overall Officials: Gethin H Evans, PhD, Principal Investigator — Manchester Metropolitan University; Adora MW Yau, PhD, Principal Investigator — Manchester Metropolitan University; John McLaughlin, Prof., Principal Investigator — University of Manchester
Locations (1):
- Manchester Metropolitan University, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Planned communication of group results at a scientific conference. Planned publication in a scientific peer reviewed journal. Participant level data is not expected to be available as this complies with the conditions of the ethical approval granted for this study.